CLINICAL TRIAL: NCT00995631
Title: Regional Fat Re-accumulation Following Lipectomy in Pre- and Post-menopausal Women
Brief Title: Following Lipectomy to Understand Adipose Tissue Re-accumulation
Acronym: FLARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 07-0339; NIH DK077992
Record Dates: First submitted 2009-10-12; First posted 2009-10-15 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Menopause; Pre-menopause
Keywords: liposuction; adipose tissue; dietary fatty acids; triglyceride storage; Normal healthy aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Premenopausal, Control (No Intervention): Premenopausal women randomized to Control (delayed liposuction surgery)
- Premenopausal, Surgery (Active Comparator): Premenopausal women randomized to surgery (femoral lipectomy)
  Interventions: Procedure: Femoral lipectomy
- Postmenopausal, Control (No Intervention): Postmenopausal women randomized to Control (delayed liposuction surgery)
- Postmenopausal, Surgery (Active Comparator): Postmenopausal women randomized to surgery (femoral lipectomy)
  Interventions: Procedure: Femoral lipectomy

INTERVENTIONS:
Procedure: Femoral lipectomy — Standard (non-experimental) suction assisted liposuction surgery
  Arms: Postmenopausal, Surgery; Premenopausal, Surgery

SUMMARY:
The typical female pattern of accumulating fat in the hips and thighs has long been thought to confer less risk for disease than the typical male abdominal fat pattern. However, leg fat may not simply be benign with respect to disease risk, but may in fact protect against cardiovascular disease risk. Although the mechanism for this is unknown, the investigators hypothesize that removing a portion of this important fat depot (via liposuction) could increase disease risk. Such unfavorable results may or may not be transient depending on an individual's ability to defend their fat mass. Because sex hormones appear to play a role in regional fat accumulation, the investigators hypothesize that estrogen-deficient postmenopausal women may have an augmented abdominal fat accumulation and an attenuated hip and thigh re-accumulation compared to premenopausal women following lipectomy and compared to non-surgical controls. As a result, the increased abdominal fat accumulation may worsen disease risk in postmenopausal women. Menopause-related differences in fat storage at baseline are also expected to determine the degree to which lipectomy alters disease risk and the propensity for AT re-accumulation.

DETAILED DESCRIPTION:
Lipectomy is the most frequently performed aesthetic surgery in the U.S. today and is considered permanent, by The American Society for Aesthetic Plastic Surgery, but no long term follow-up studies have been done to verify this assertion. Indeed, animal studies suggest rapid adipose tissue (AT) re-accumulation after lipectomy is common and may even be accompanied by unfavorable changes in disease risk. Recent studies in humans have focused on abdominal lipectomy as a means of reducing metabolic disease risk in obese premenopausal women. However, none of these studies evaluated AT re-accumulation or reported long-term (>6 mo) changes in metabolic outcomes, and none have evaluated the effect of removing femoral AT despite this being a common site for lipectomy in women and despite the apparent cardioprotective benefit of lower body adiposity. Further, none of these studies included postmenopausal women who are at an increased risk of abdominal AT accumulation. It is the investigator's overall working hypothesis that removal of femoral AT by lipectomy may worsen metabolic disease risk (as measured by postprandial lipemia) in estrogen-deficient postmenopausal women who, in contrast to premenopausal women, will accumulate AT in the abdominal rather than the femoral region. The global aims of this study are to determine whether: 1) there are menopause-related differences in regional (abdominal vs. femoral) AT re-accumulation following lipectomy; and 2) changes (removal and regain) in femoral AT mass alter postprandial triglyceride clearance and storage of meal-derived fatty acids. Further, the investigators postulate that menopause-related differences in postprandial lipemia and handling of dietary fatty acids will determine the degree to which femoral lipectomy worsens these parameters. Pre- and postmenopausal women (n=80) will be randomly assigned to either femoral lipectomy or control (no surgery). All eligible volunteers will undergo testing at the beginning of the study and at 2, 8, and 14 months following lipectomy. Measurements will include body composition assessments, meal tests and AT biopsies to assess lipectomy-related changes in: 1) abdominal and femoral fat mass; 2) systemic postprandial triglyceride excursions; and 3) storage of dietary fatty acids in AT. These studies are designed to evaluate the effect of femoral lipectomy on regional AT re-accumulation and metabolic disease risk in pre- and postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal (no menses for 12mo or oophorectomy w/ follicle-stimulating hormone (FSH)>30 IU/L) OR- pre-menopausal (regular menses 28+/-3d)
* BMI >20 and <30 kg/m2)
* weight stable (+/- 2kg in past 2mo)
* non-smoking
* no use of hormone therapies or oral contraceptives
* actively seeking liposuction of the hips and thighs
* good femoral lipectomy candidates as determined by cosmetic surgeon

Exclusion Criteria:

* severe hypertriglyceridemia (>400 mg/dL)
* medications known to affect lipid metabolism
* elevated resting blood pressure (Systolic >140 mm Hg,Diastolic >90 mm Hg)
* history of lipectomy or gastric bypass surgery
* body dysmorphic disorder
* pregnant, lactating or intention of becoming pregnant
* indication of high surgical risk (e.g., abnormal resting ECG, history of thromboembolism, valvular heart disease)

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2008-01; Primary Completion 2013-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postprandial triglyceride excursions (incremental areas) | Baseline, 2Mo, and 14Mo
Abdominal and femoral fat mass accumulation | Baseline, 2Mo, and 14Mo

SECONDARY OUTCOMES:
Triglyceride storage (14C-oleic acid incorporation into abdominal and femoral adipose tissue) | Baseline, 2Mo, and 14Mo
Lipoprotein lipase activity (abdominal and femoral adipose tissue) | Baseline, 2Mo, and 14Mo

CONTACTS AND LOCATIONS:
Overall Officials: Rachael E Van Pelt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States